CLINICAL TRIAL: NCT06349122
Title: Screen-and-treat Strategy for Vaginal Flora Abnormalities by Multiplex Molecular Biology Using POC Technology in Pregnant Women at High Risk of Preterm Birth: A Multicentre, Randomized Study (AUTOP2)
Brief Title: Screen-and-treat Strategy for Vaginal Flora Abnormalities in Pregnant Women at High Risk of Preterm Birth
Acronym: AUTOP2
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-509421-41-00
Record Dates: First submitted 2024-03-14; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Bacterial Vaginosis; Vaginal Dysbiosis; Premature Delivery
Keywords: screen and treat strategy
MeSH Terms: conditions — Vaginosis, Bacterial; Premature Birth | interventions — Azithromycin; Ceftriaxone; Metronidazole; Clotrimazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Screen-and-Treat Strategy (Experimental): Patients are systematically screened for BV before 18 weeks' gestation by means of a vaginal swab analyzed by the innovative technique, whose result will be disclosed. If positive, appropriate treatment will be prescribed.
  Interventions: Diagnostic Test: Vaginal flora abnormalities screening and quantification using molecular biology technique; Drug: Azithromycine; Drug: Ceftriaxone; Drug: Metronidazole; Drug: Clotrimazole, Vaginal
- Group B: Control Group/Usual Care or Standard Strategy (Active Comparator): Patients are not systematically screened for BV /usual care group.
  Interventions: Other: Usual Care

INTERVENTIONS:
Diagnostic Test: Vaginal flora abnormalities screening and quantification using molecular biology technique — Vaginal self-sampling is a simple and validated method of sampling used for the molecular biology technique and the quantification of microorganisms involved in vaginal flora imbalance bacteriosis.The patient performs a self-sampling with a cotton swab transferred into a transport medium tube. The sample is sent to the laboratory where Multiplex Point of Care polymerase chain reaction (PCR) is performed.
  Arms: Group A: Screen-and-Treat Strategy
Drug: Azithromycine — In case of Chlamydia trachomatis infections, as well as significant increase of Fannyhessea vaginae: 1 g per os in a single dose; In case of Neisseria gonorrhoeae infection: 2 g per os in a single dose (associated to ceftriaxone 1g IM)
  Arms: Group A: Screen-and-Treat Strategy
Drug: Ceftriaxone — In case of Neisseria gonorrhoeae infections, 1g, associated to azithromycin 2 g per os in a single dose
  Arms: Group A: Screen-and-Treat Strategy
Drug: Metronidazole — Metronidazole ovules: In case of Trichomonas vaginalis infection during the 1st trimester of pregnancy: 1 ovule morning and evening for 14 days (French Society of Dermatology Recommendations 2016); Metronidazole 500 mg tablets in case of Trichomonas vaginalis infection during the 2nd or the 3rd trimester of pregnancy in a single dose of 2 g
  Arms: Group A: Screen-and-Treat Strategy
Drug: Clotrimazole, Vaginal — In case of Candida albicans infection in a single dose to be repeated up to 6 times if necessary.
  Arms: Group A: Screen-and-Treat Strategy
Other: Usual Care — Patients will not be screened using molecular biology techniques in this group. The management of these patients is a matter of routine for health professionals. They will be free to prescribe a standard vaginal swab if symptoms are present and to treat their patients according to their usual protocols. No routine sampling is recommended in the absence of a history
  Arms: Group B: Control Group/Usual Care or Standard Strategy

SUMMARY:
Preterm birth is an important cause of death and disabilities. Bacterial vaginosis (BV) is a common vaginal dysbiosis or abnormal microbiota, with a predominance of anaerobic bacteria with a lack of Lactobacillus, with various diagnosis methods. Often asymptomatic, BV increases the risk of preterm birth according to the gestational age at diagnosis. BV is usually diagnosed by conventional diagnosis such as Nugent score. Molecular diagnosis of BV has been demonstrated to be more reproducible, more accurate and to better define dysbiosis.

The main objective of the study is to evaluate the effectiveness of an innovative screen-and-treat strategy for vaginal flora abnormalities by molecular biology using a Point of Care multiplex technology before 18 weeks' gestation to reduce the rate of preterm birth in a population of pregnant women at high risk of preterm birth.

The hypothesis is that a strategy for screening and treating vaginal flora abnormalities and their recurrences using molecular biology in women with a history of prematurity or late-term abortion could be effective in reducing premature births by 40%.

DETAILED DESCRIPTION:
Preterm birth is an important cause of death and disabilities. Bacterial vaginosis (BV) is a common vaginal dysbiosis or abnormal microbiota, with a predominance of anaerobic bacteria with a lack of Lactobacillus with various diagnosis methods. Often asymptomatic, BV increases the risk of preterm birth according to the gestational age at diagnosis. BV is usually diagnosed by conventional diagnosis such as Nugent score. Molecular diagnosis of BV has been demonstrated to be more reproducible, accurate and to better define dysbiosis.

AUTOP was a large randomized multicentre trial to evaluate a "Screen and Treat" strategy for bacterial vaginosis using molecular diagnosis of self-collected vaginal samples in low-risk pregnant women during early pregnancy, with an evaluation of treatment success, and including vaginal swab controls.

Among 6,671 randomized women, the Intent to treat analysis of the primary clinical outcome showed no evidence of a reduction in the rate of preterm birth with the screen and treat strategy compared with usual care. The rate of preterm birth was 3.9% (events=127) among 3,333 women in the screen and treat strategy group and 4.6% (events=153) among 3,338 in the control group (aOR, 0.82 [95%CI, 0.65 to 1.05]; P=.12). In the subgroup of nulliparous women (n=3,438), Screening and treating strategy was significantly more effective than usual care (aOR 0.61, 95% CI 0.44 to 0.82; Pinteraction=0.001).

AUTOP I has been submit to JAMA at the beginning of 2023. AUTOP was the first randomized study that evaluates the impact of Screen and Treat strategies using molecular biology during pregnancy, except one ongoing study.

The main objective of AUTOP 2 study is to evaluate the effectiveness of an innovative screen-and-treat strategy for vaginal flora abnormalities by molecular biology using Point of Care multiplex technology before 18 weeks' gestation to reduce the rate of preterm birth in a population of pregnant women at high risk of preterm birth (with previous history of preterm birth or late fetal loss) , in comparison with a standard strategy with absence of screening.

AUTOP 2 is a multicenter, prospective, randomized, parallel, open-label comparative study comparing 2 groups of pregnancy management in a population of pregnant women at high risk of preterm birth.

* Screen-and-Treat Innovative Strategy (Group A): patients systematically screened for BV before 18 weeks of gestation by means of a vaginal swab analyzed by the innovative technique, whose result will be disclosed. If positive, appropriate treatment will be prescribed.
* Control Group/Usual Care or Standard Strategy (Group B): patients not systematically screened for BV/usual care group.

The recruitment goal is of 1292 women (646 per group). The period of inclusion has been scheduled to be 24 months. Each subject will be followed for a period of 17 months (maximum 7 months of pregnancy until term and 10 months post-delivery).

A reduction in prematurity and/or late abortions in the group screening and treatment of vaginal flora abnormalities is expected. This strategy could be implemented routinely if the results were significant.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women over 18 years of age
* Pregnant woman after 8 weeks and before 18 weeks of gestation (i.e. >=8 weeks and ≤ 18 weeks)
* Woman who has understood the study process and objectives and agreed to sign an informed consent form;
* With a history of preterm birth before 37 weeks of gestation or late miscarriage (high-risk preterm birth population) (A late miscarriage or late fetal loss mean foetal loss between 14 and 22 weeks of gestation)
* Affiliated to a social security regimen or equivalent

Exclusion Criteria:

* - Woman of legal age under legal protection;
* Women deprived of their freedom for administrative or legal reasons;
* Woman who has not signed a consent form
* Nulliparous;
* Ectopic pregnancy;
* Non-evolutive pregnancy or IUFD
* Multiple pregnancy
* Serious fetal malformation identified at first trimester screening such as cardiopathy, exencephaly, anasarque, gastroschisis, omphalocele, diaphragmatic hernia, cerebral or spinal major anomaly.
* Woman participating in any clinical trial or intent to participate in another clinical trial, which may have an impact on flora or on prematurity rate, with or without investigational product at any time during the conduct of this study
* Woman presenting contraindications to the study treatments: Hypersensitivity to the active substance or to any of the excipients
* Woman presenting uterine malformation ( unicornuate, bicornuate, full septate)
* Woman with preterm birth history because of twin pregnancy
* Woman having received anti-infective treatment in the week preceding inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women at high risk of preterm birth
Enrollment: 1292 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
The rate of preterm birth | Before 37 weeks of gestation
  The primary endpoint will be the rate of preterm birth before 37 weeks of gestation, which will be compared between the innovative group and the standard group.

IPD SHARING:
Plan to Share IPD: No